CLINICAL TRIAL: NCT05572788
Title: Randomized Trial of Rectal Indomethacin to Prevent Acute Pancreatitis in Patients Undergoing Endoscopic Ultrasound-guided Fine Needle Aspiration of Pancreatic Cysts
Brief Title: Rectal Indomethacin to Prevent Acute Pancreatitis in EUS-FNA of Pancreatic Cysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 22.085.04; 1894054 (Other: Orlando Health IRB)
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cyst; Pancreatitis, Acute
MeSH Terms: conditions — Pancreatic Cyst; Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rectal Indomethacin (Active Comparator): Patients assigned to the Indomethacin group will receive100 mg of indomethacin administered per rectal route (two tablets of 50 mg indomethacin suppositories)
  Interventions: Procedure: EUS-guided fine needle aspiration of pancreatic cysts
- Placebo (Placebo Comparator): Patients assigned to the Placebo group will receive two glycerin suppositories.
  Interventions: Procedure: EUS-guided fine needle aspiration of pancreatic cysts

INTERVENTIONS:
Procedure: EUS-guided fine needle aspiration of pancreatic cysts — Patients with pancreatic cysts requiring fine needle aspiration will be enrolled in this randomized trial

SUMMARY:
The aim of this randomized trial is to compare the rate of post-procedure pancreatitis in patients undergoing EUS-FNA of pancreatic cysts; patients will receive either a single dose of indomethacin or placebo administered rectally, during EUS-FNA.

DETAILED DESCRIPTION:
Pancreatic cysts are pre-malignant lesions and are being increasingly diagnosed on cross-sectional imaging. Endoscopic ultrasound (EUS) is performed to further evaluate pancreatic cysts, and fine needle aspiration (FNA) is conducted to obtain a sample of the cystic fluid for analysis and examination for malignant cells. Acute pancreatitis is a complication of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) of pancreatic cysts, which can lead to significant morbidity and substantial health care costs. The aim of this randomized trial is to compare the rate of post-procedure pancreatitis in patients undergoing EUS-FNA of pancreatic cysts; patients will receive either a single dose of indomethacin or placebo administered rectally, during EUS-FNA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suspected or confirmed pancreatic cyst seen on imaging, requiring EUS-FNA

Exclusion Criteria:

* Unable to obtain consent from the participant or the participant's legally authorized representative (LAR)
* Intrauterine pregnancy
* Hypersensitivity reaction to Aspirin or NSAIDs
* Patients with known history of chronic pancreatitis
* Patients with known renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of post-procedure pancreatitis following EUS-guided fine needle aspiration of pancreatic cysts | 30 days
  Post-procedure pancreatitis is defined as the development of new or increased abdominal pain consistent with acute pancreatitis, and elevated amylase or lipase at least three times the upper limit of normal .

SECONDARY OUTCOMES:
Rate of procedure-related adverse events | 30 days
  Rate of adverse events resulting from EUS-FNA
Disease-related adverse events | 30 days
  Any adverse event occurring as a result of underlying pancreatic cyst
Rate of mild, moderate and severe pancreatitis post-FNA | 30 days
  Rate of mild, moderate and severe pancreatitis post-FNA
Length of hospitalization in any patient hospitalized with any adverse event | 30 days
  Length of hospitalization in any patient hospitalized with any adverse event
Length of hospitalization in any patient hospitalized with acute pancreatitis | 30 days
  Length of hospitalization in any patient hospitalized with acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health, Digestive Health Institute
Locations (1):
- Orlando Health, Orlando, Florida, United States